CLINICAL TRIAL: NCT03107728
Title: The IM ABLE Study: A Cross-Sector, Multisite Initiative to Advance Care for Warriors and Veterans Following Neuromusculoskeletal Injury of the Lower Limb
Brief Title: The IM ABLE Study: A Study of Warriors & Veterans Following Neuromusculoskeletal Injury of the Lower Limb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: James A. Haley Veterans Administration Hospital (U.S. Federal Agency); VA New York Harbor Healthcare System (U.S. Federal Agency); Hanger Clinic: Prosthetics & Orthotics (Other)
Responsible Party: Principal Investigator, Jason Highsmith, Associate Professor, University of South Florida
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00026645; W81XWH-16-1-0738 (Other Grant/Funding Number: USAMRAA)
Record Dates: First submitted 2017-03-29; First posted 2017-04-11 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Limb Salvage; Braces; Lower Extremity
Keywords: orthotics; high-energy lower extremity trauma; physical therapy; bracing; functional performance; performance assessment

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced orthotic brace (Experimental)
  Interventions: Device: Advanced orthotic brace
- Conventional orthotic brace (Active Comparator)
  Interventions: Device: Conventional orthotic brace

INTERVENTIONS:
Device: Advanced orthotic brace — Participants will use an advanced exoskeletal orthosis.
  Arms: Advanced orthotic brace
Device: Conventional orthotic brace — Participants will use the standard of care orthosis
  Arms: Conventional orthotic brace

SUMMARY:
The purpose of the IM ABLE(Injuries Managed with Advanced Bracing for Lower Extremities) study is to determine if advanced (ADV) ankle foot orthoses (AFOs) will enable users to achieve greater levels of physical and self-reported function compared with conventional (CONV) AFOs for those ambulating at or above the independent community level of ambulation.

DETAILED DESCRIPTION:
There were approximately 20,000 extremity trauma cases associated with the wars in Iraq and Afghanistan. Many of these individuals have experienced multiple limb-sparing surgeries and orthotic utilization. Many continue functioning with use of their orthosis while others may seek delayed amputation. It is unclear if limb salvage or amputation is more advantageous functionally or preferred following lower extremity(LE) trauma. The IDEO (Intrepid Dynamic Exoskeletal Orthosis) was developed to assist in maintaining high functional performance in patients who have experienced high energy lower extremity trauma (HELET) and limb salvage surgeries primarily effecting the LE below the level of the knee joint. The IDEO represents one "advanced" orthotic option for a traumatized and surgically spared limb however there are other "advanced" orthotic options. Problematically, few studies have reported outcomes associated with these devices. In the few studies available, sample sizes are small which greatly reduces generalizability of study findings. The purpose of the IM ABLE study is to determine if advanced (ADV) ankle foot orthoses (AFOs) will enable users to achieve greater levels of physical and self-reported function compared with conventional (CONV) AFOs for those ambulating at or above the independent community level of ambulation.

ELIGIBILITY:
Inclusion Criteria:

1. Lower extremity injury of any etiology requiring use of an AFO
2. Male or Female, of any ethnicity
3. 18-65 yrs of age
4. 100-275 lbs
5. ≥ 1 yr. of orthotic experience

Exclusion Criteria:

1. Body weight <100 or >275 lbs
2. Does not speak English or Spanish
3. Known cognitive impairment (i.e. Diagnoses such as Traumatic Brain Injury, Dementia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change in Mobility | Mobility will be assessed at Week 2 and Week 4
  Mobility will be assessed with the Timed Up & Go test. subjects are timed while they rise from a chair, walk 3m, turn around, return to the chair and sit down again. Patients are usually permitted to use a walking aid, but not to use physical assistance.
Change in Ambulatory Function | Ambulatory Function will be assessed at week 2 and week 4.
  The 2 Minute Walk Test will be used to assess ambulatory function

SECONDARY OUTCOMES:
Perceived Function | At week 2 and week 4
  Perceived Function will be assessed via the EQ-5D (EuroQol 5D), a five item ordinally scaled patient self-report.
Pain | At week 2 and week 4
  Pain rating scale 0-10
Safety will be measured with the Activities Balance Confidence Scale | At week 2 and week 4
  Safety will be measured with the Activities Balance Confidence Scale, a 16 item self-report measure of perceived balance confidence

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - New York VA, New York, New York
  - Hanger, Inc, Houston, Texas